CLINICAL TRIAL: NCT06867276
Title: Low Level Laser Versus Polarized Light in the Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sohila Mamdouh Morsy Mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sohaila-004677
Record Dates: First submitted 2025-02-28; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Low Level Laser Therapy; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Lasers, Excimer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Excimer laser (Experimental): This group includes 25 patients; all the participants received low level laser (Excimer laser) in a series of eight treatment sessions that was performed twice per week. The radiation exposure time is 10 minutes during the procedure, a maximum dose of 0.65 J/cm², and 6 different spot sizes to avoid healthy skin. large spot size (20 cm²).
  Interventions: Device: Excimer laser
- Bioptron (Active Comparator): This group includes 25 patients; all the participants received polarized light (Bioptron Pro l) in a series of eight treatment sessions that was performed twice per week. The radiation exposure time is 10 minutes during the procedure; a device is fixed at a distance of 10 cm from the treatment area (face), light spot size 19 cm2 average power density is 40 mille watt per cm², and a dose of 2.4 J/cm² per minute.
  Interventions: Device: Bioptron Pro 1

INTERVENTIONS:
Device: Excimer laser — Excimer laser patients undergo ultraviolet b phototherapy treatments at a physical medicine clinic twice a week for four weeks. The device uses a 308nm beam of coherent light, with six spot sizes to avoid healthy skin. The radiation exposure time is 10 minutes, with a maximum dose of 0.65 J/cm². Personal protection standards include wearing protective eyewear for the retina and choroid, as they absorb visible light radiation, which can cause keratoconjunctivitis or cataracts. The thermal effect of the laser can cause superficial carbonization of the epidermis, phlyctens, or erythema, so non-flammable gloves are recommended.
  Arms: Excimer laser
Device: Bioptron Pro 1 — Patients undergone Bioptron light treatment twice weekly for four weeks at a physical medicine clinic. The treatment is administered by a physiatrist following the manufacturer's user guide. Patients sit in a comfortable chair with their hand on an armrest, holding the Bioptron light probe at a 90° angle for 10 minutes.
  Arms: Bioptron

SUMMARY:
The present study is designed to compare clinically the therapeutic applications between low level laser therapy (excimer laser) and non-laser polarized light (Bioptron prol) in the treatment of Acne vulgaris.

DETAILED DESCRIPTION:
Traditional acne treatment often involves topical application, which can cause skin irritation and dryness, and oral antibiotic therapy, which is limited by antibiotic resistance. Newer procedures like laser and light-based therapies offer alternative treatments for patients who struggle with adherence or experience side effects or treatment failure. This study aims to compare the therapeutic application of laser and light therapies as an alternative to traditional acne treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients.
2. Age range between 18 and 25 years.
3. All patients will sign their informed consent to participate in the research procedure and to publish the data.
4. Definite clinical diagnosis of mild to moderate inflammatory lesions of facial Acne vulgaris (open and closed comedones, papules, pustules, and nodules) on the face that has been going on for at least 1 month.

Exclusion Criteria:

1. Patient's unwillingness to continue cooperation in the study
2. Photosensitive skin.
3. Pregnancy and breast feeding.
4. Women who use hormonal contraceptives.
5. Patients who had used oral retinoids or any other treatment for acne in the last month.
6. Patients with severe nodulocystic acne

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
assessment of change of Global Assessment Scale | At baseline and after 4 weeks
  For the study, we recruited males and females with mild to moderate acne according to the Investigator's Global Assessment (IGA) scale, where the severity of acne and the type of lesions was assigned to it.
  the scoring ranges from 0 to 4. Zero indicates clear skin with no inflammatory and non- inflammatory lesions, while 4 indicates severe lesion with Many comedones and inflammatory lesions, ≤ several nodules and cysts

SECONDARY OUTCOMES:
assesment of change of digital facial photographs | At baseline and after 4 weeks
  Digital Facial photographs, included in the photographic documentation, were taken by (Nikon Camera), before the procedure and four weeks after the end of the whole therapy.
  Digital facial photographs will be taken for each patient at the base line and end of the fourth week to track the development of acne lesions and evaluate treatment effectiveness, using the same method for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No